CLINICAL TRIAL: NCT06783868
Title: Randomized Control Study to Assess the Neurological Outcomes After Atrial Fibrillation Ablation for Rhythm Control vs Routine Medication Therapy in Patients With Recent Stroke: SAVE STROKE Phase II Study
Brief Title: Assessing the Neurological Outcomes After Atrial Fibrillation Ablation for Rhythm Control
Acronym: SAVE STROKE II
Status: Not yet recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_SAVE STROKE II_0037
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Routine Medication Therapy: Will receive SOC following AF diagnosis in the setting of stroke. This includes rate control with a combination of atrioventricular nodal blockers (AVNB) (Metoprolol, Diltiazem, etc.) and initiation of oral anticoagulation (OAC) (either Eliquis, Xarelto, or Warfarin) within 1-14 days per recommendations of the Stroke Team. If arrhythmia remains uncontrolled, patients will be started on an anti-arrhythmic drugs (AAD) (either Flecainide, Dofetilide, Propafenone, Sotalol, Amiodarone, etc.) per Electrophysiology. Doses of medications will be determined by the managing physician. If a patient was/is started or on triple therapy, this will be converted to appropriate anti-platelet and OAC. Patients will continue this management if AF is controlled. Patients can still undergo CA for rhythm control at the discretion of the managing Electrophysiologist.
  Interventions: Drug: Market-approved AVNB, OAC and AAD
- Atrial Fibrillation Ablation: When randomized to this group, patients will subsequently receive earlier rhythm control. They will undergo SOC following AF diagnosis in the setting of stroke as above. This can include AVNB and OAC. However, these patients will also be assigned to start AAD before discharge from the hospital. They will subsequently undergo CA 30-120 days from discharge from the hospital. The lesions to be ablated will be determined by electrophysiology study (EPS) with electroanatomic mapping and subsequently selected by the operator to optimize each patient situation.
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Catheter Ablation — Catheter Ablation is commonly performed with radiofrequency or cryotherapy to maintain a rhythm control strategy if patients can no longer tolerate their symptoms or are no longer controlled on AVNB or AAD. The procedure leads to significant symptom improvement even though there may be insignificant AF recurrence at one year. At Kansas City Heart Rhythm Institute, CA may be performed with radiofrequency ablation (Tactiflex Ablation Catheter, Abbott Cardiovascular, Minneapolis, MN) or pulsed field ablation (PulseSelectTM, Abbott Cardiovascular or FaraWaveTM, Boston Scientific, Marlborough, MA), performed with EnsiteX (Abbott Cardiovascular) or Carto3 (Biosense Webster, Irvine, CA) mapping software.
  Groups: Atrial Fibrillation Ablation
Drug: Market-approved AVNB, OAC and AAD — Used per protocol for the duration of the trial.
  Groups: Routine Medication Therapy

SUMMARY:
A prospective, non-blinded, multi-center study to assess the impact of early Catheter Ablation (CA) in patients with a new diagnosis of Atrial Fibrillation(AF) at the time of stroke. 100 patients will be enrolled.

DETAILED DESCRIPTION:
A prospective, non-blinded, multi-center study to assess the impact of early CA in patients with a new diagnosis of AF at the time of stroke. At least 100 patients who meet the inclusion and exclusion criteria will be randomized 1:1 to receive early CA or SOC (Standard of Care). The primary outcome will be the functional neurologic outcomes, including mRS (modified Rankin Scale) and QOL(Quality of Life), recurrence, major bleeding, and mortality after stroke for each group. Secondary outcomes will be changes in cognitive assessment, success of rhythm control, recurrent hospitalizations, and cumulative cardiovascular outcomes. Participants will be followed at 3, 6, 9, and 12 months following the discharge date to measure these outcomes, and the study will enroll for one year. The primary endpoints will be functional recovery and enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Ages >18 and able to provide consent.
* Presenting with an acute stroke and new-onset AF
* Modified RANKIN score (mRS) < 6
* Must be able to undergo some form of cardiac monitoring [implantable loop recorder (ILR), electrocardiogram (ECG), Holter monitor] to quantify AF burden

Exclusion Criteria:

* Patients < 18 years of age
* Unable to provide consent, including mRS = 6.
* Not able to read and write at an 8th-grade level [to complete AFEQT and EQ-5D surveys]
* Positive B-hCG
* Will not follow up with our practice/clinic afterward.
* Cannot tolerate OAC or AAD for any reason.
* Cannot undergo CA for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation (AF) and recent stroke.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Functional neurologic outcome - Modified Rankin Scale | 1 Month, 3 Months, 6 Months, 9 Months and 12 Months
  Modified Rankin Scale is widely used to assess neurologic dysfunction in a broad range of neurologic and neurosurgical conditions. It is a 6-level ordinal outcome scale (0-5) used to assess the functional status of patients, encoding the range from no symptoms or functional impairment (mRS = 0) to severe disability requiring constant nursing care (mRS = 5)
Recurrent Stroke | 12 Months
  A recurrent stroke is when a person has another stroke following their first stroke. Experiencing one can have a major impact on a person's quality of life.

SECONDARY OUTCOMES:
Functional neurologic outcome - Quality of Life | 1 Month, 3 Months, 6 Months, 9 Months and 12 Months
  The AF Effect on Quality-of-Life questionnaire - AFEQT for short - is a reliable and responsive measure of quality of life, developed especially for atrial fibrillation. Overall or subscale scores range from 0-100.
  A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (7):
- United States (7):
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] About Stroke. 2023
- [Background] What is Atrial Fibrillation.2023
- [Background] Roman S, Patel K, Hana D, Guice KC, Patel J, Stadnick C, Basta A, Khouzam RN. Rate versus rhythm control for atrial fibrillation: from AFFIRM to EAST-AFNET 4 - a paradigm shift. Future Cardiol. 2022 Apr;18(4):354-353. doi: 10.2217/fca-2021-0034. Epub 2022 Mar 8. PMID 35255732
- [Background] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbuchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 1;383(14):1305-1316. doi: 10.1056/NEJMoa2019422. Epub 2020 Aug 29. PMID 32865375
- [Background] Bunch TJ, Crandall BG, Weiss JP, May HT, Bair TL, Osborn JS, Anderson JL, Muhlestein JB, Horne BD, Lappe DL, Day JD. Patients treated with catheter ablation for atrial fibrillation have long-term rates of death, stroke, and dementia similar to patients without atrial fibrillation. J Cardiovasc Electrophysiol. 2011 Aug;22(8):839-45. doi: 10.1111/j.1540-8167.2011.02035.x. Epub 2011 Mar 15. PMID 21410581
- [Background] Park J, Shim J, Lee JM, Park JK, Heo J, Chang Y, Song TJ, Kim DH, Lee HA, Yu HT, Kim TH, Uhm JS, Kim YD, Nam HS, Joung B, Lee MH, Heo JH, Pak HN; RAFAS Investigators*. Risks and Benefits of Early Rhythm Control in Patients With Acute Strokes and Atrial Fibrillation: A Multicenter, Prospective, Randomized Study (the RAFAS Trial). J Am Heart Assoc. 2022 Feb;11(3):e023391. doi: 10.1161/JAHA.121.023391. Epub 2022 Jan 19. PMID 35043663
- [Background] Jensen M, Suling A, Metzner A, Schnabel RB, Borof K, Goette A, Haeusler KG, Zapf A, Wegscheider K, Fabritz L, Diener HC, Thomalla G, Kirchhof P. Early rhythm-control therapy for atrial fibrillation in patients with a history of stroke: a subgroup analysis of the EAST-AFNET 4 trial. Lancet Neurol. 2023 Jan;22(1):45-54. doi: 10.1016/S1474-4422(22)00436-7. PMID 36517170
- [Background] Turagam MK, Musikantow D, Whang W, Koruth JS, Miller MA, Langan MN, Sofi A, Choudry S, Dukkipati SR, Reddy VY. Assessment of Catheter Ablation or Antiarrhythmic Drugs for First-line Therapy of Atrial Fibrillation: A Meta-analysis of Randomized Clinical Trials. JAMA Cardiol. 2021 Jun 1;6(6):697-705. doi: 10.1001/jamacardio.2021.0852. PMID 33909022